CLINICAL TRIAL: NCT02590536
Title: A Randomized Controlled Trial Evaluating the Role of Sildenafil in the Treatment of Fetal Growth Restriction
Brief Title: A Trial Evaluating the Role of Sildenafil in the Treatment of Fetal Growth Restriction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFGR
Record Dates: First submitted 2015-10-21; First posted 2015-10-29 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Fetal Growth Retardation
Keywords: Sildenafil; Fetal growth Restriction; Umbilical Artery Doppler
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- sildenafil citrate (Experimental): Group A (45 patients): pregnancies affected by Fetal Growth Restriction (FGR) being treated with sildenafil citrate 25 mg of sildenafil citrate every 8 hours starting at diagnosis of FGR until delivery
  Interventions: Drug: Sildenafil citrate
- placebo (Placebo Comparator): Group B (45 patients): pregnancies affected by Fetal Growth Restriction (FGR) being treated with placebo every 8 hours starting at diagnosis of FGR until delivery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sildenafil citrate — In patients with Fetal Growth Restriction (FGR)and abnormal umbilical artery Doppler, will be randomly assigned and divided to 2 groups which will be treated with sildenafil citrate either placebo.
  This study will compare the change in Resistance Index (RI) and the Pulsatility Index (PI) of the umbilical artery and fetal middle cerebral artery, for patients who receive 25 mg of oral sildenafil citrate 8 hourly starting at diagnosis of FGR until delivery against those who will receive placebo of the same color and shape of sildenafil citrate tablet.
  Arms: sildenafil citrate
Drug: placebo
  Arms: placebo

SUMMARY:
This is a Randomized Controlled Trial to evaluate the effect of sildenafil on Doppler velocity indices of the umbilical arteries in patients with placental insufficiency and fetal growth restriction, and if sildenafil can improve fetal and neonatal outcomes in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, singleton pregnancy, gestational age 24-34 weeks, with

  * Fetal growth restriction.
  * Intact membranes.
  * Abnormal umbilical artery Doppler waveforms.
* Fetal abdominal circumference at or below the tenth percentile.
* Normal venous fetal Doppler

Exclusion Criteria:

* Undetermined gestational age.
* Intrauterine infection.
* High Risk for aneuploidy (e.g. maternal age ≥40 years, detected congenital fetal anomalies in the current or previous pregnancies).
* Maternal cardiovascular morbidity.
* Users of any vasodilator agents.
* Known allergy to sildenafil citrate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
The change in Doppler velocity indices( Resistance index (RI) and the pulsatility index (PI) of the umbilical arteries as a Ratio | 24 weeks to 34 weeks of gestation.
The change in Doppler velocity indices( Resistance index (RI) and the pulsatility index (PI), of fetal middle cerebral artery as a Ratio | 24 weeks to 34 weeks of gestation.

SECONDARY OUTCOMES:
Neonatal birth weight in grams | At time of Delivery
Gestational age at delivery in weeks | At time of Delivery
Neonatal complication rates including Intraventricular hemorrhage (IVH) , Neonatal Necrotizing Enterocolitis (NEC) , Syndrome Respiratory Distress (RDS) , Neonatal anemia, Neonatal blood transfusion). | The first 28 day of delivery
Neonatal ICU admission rate | The first 28 day of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Khaled I Abdullah, MD, Study Chair — Ain Shams University; Sherif A Ashoush, MD, Principal Investigator — Ain Shams University; Heba E Hosney, MSc, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt